CLINICAL TRIAL: NCT06687603
Title: Multi-Site Detection of Barrett's Esophagus in Patients Without Chronic GERD Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASE10224
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux; Esophageal Adenocarcinoma
Keywords: Esophagus; Non-endoscopic
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Masking Description: All endoscopic images will be reviewed by an examiner who will be blinded to the endoscopy report. BE will be defined as the presence of > 1 cm of columnar appearing epithelium in the tubular esophagus as confirmed by the blinded reviewer plus the presence of intestinal metaplasia on biopsies. I
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EsoCheck + EsoGuard (Experimental): Participants will undergo an EsoCheck test. The sample produced by the EsoCheck will be sent to LucidDx where the EsoGuard assay will be performed.
  Interventions: Device: EsoCheck; Diagnostic Test: EsoGuard

INTERVENTIONS:
Device: EsoCheck — FDA-approved, non-endoscopic, encapsulated swallowable balloon. EsoCheck will produce a sample which will subsequently be tested with EsoGuard assay. The EsoCheck is performed and completed in approximately 5 minutes.
Diagnostic Test: EsoGuard — Approved laboratory, methylated DNA panel that detects esophageal neoplasia. The EsoGuard assay tests the EsoCheck samples to detect BE in GERD participants.

SUMMARY:
The goal of this clinical trial is to develop a method to detect Barrett's esophagus in individuals with a new office based diagnostic test. Barrett's esophagus is a condition in which the flat pink lining of the swallowing tube that connects the mouth to the stomach (the esophagus) becomes damaged by acid reflux. The main question it aims to answer is: Can this approach demonstrate efficacy for screening of Barrett's esophagus?

Participants will:

* Participate in a questionnaire.
* Undergo a capsule balloon test, called EsoCheck.
* Have their EsoCheck sample sent to the laboratory for an EsoGuard test, which is used to detect Barrett's esophagus.
* Participants will undergo upper endoscopy as part of standard of care.

DETAILED DESCRIPTION:
The overall goal of this clinical trial is to eliminate deaths from Esophageal Adenocarcinoma (EAC) by demonstrating the efficacy of a non-endoscopic method for efficient population screening to detect all Barrett's esophagus (BE), the precursor lesion of EAC. EAC is a highly lethal malignancy with less than 20% 5-year survival, and an annual U.S. incidence > 14,000 that has increased more than 6-fold in the past three decades. Barrett's esophagus, a pre-malignant metaplasia/neoplasia, is the precursor lesion of EAC, but is currently detectable only when patients undergo upper endoscopy (EGD). Despite Guideline recommendations for EGD in chronic GERD (gastrointestinal reflux disease) patients, barriers to EGD that include cost, sedation, and lack of acceptance, have so severely limited screening that antecedent BE remains undetected in over 95% of EAC cases. A major advance in EAC prevention was made by developing a non- endoscopic biomarker based method for detecting BE. The technology consists of an encapsulated swallowable balloon (EsoCheck) enabling a 5 minute non-endoscopic sampling of the esophagus, combined with a methylated DNA panel that detects esophageal neoplasia (EsoGuard). The research team validated the > 90% sensitivity and specificity of EC+EG testing in the population of individuals who have symptomatic GERD, and who account for 60% of EAC cases. In this new proposal, the research team plans to double the impact of this technology to detect nearly all individuals harboring BE, by proving the EC+EG technology is so robust that it further enables screening a population of high risk, but asymptomatic, non-GERD individuals who account for the remaining 40% of EAC cases, but who fall totally outside of all current screening guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing screening colonoscopy are an accessible cohort for BE screening and are also a reasonable representation of the general population. Permission will be obtained from colonoscopy physicians for researchers to contact and recruit patients for this study. Patients without GERD, who are at risk for BE, and who have not had a prior EGD, will be recruited prior to or at the time of scheduled colonoscopy.(9) Those eligible will be:

* Adults who have not had prior EGD within past ten years, and are able to provide informed consent, and who have:
* No known coagulopathy, no known esophageal varices, not on chronic anticoagulation therapy, and have:
* No significant dysphagia or odynophagia; but who do have:
* Absence of GERD (absence of weekly heartburn or regurgitation, not on medications for GERD), and are:
* Adults > age 50, who also have two or more added risk factors for BE from the set of: central obesity (waist size > 35 inches for women and > 40 inches for men), current smoker or smoking history > 10 pack years, white race, male sex, confirmed history of BE/EAC in at least two family members, with one a first degree relative. While BE is most highly prevalent in white males, a black female over age 50 with obesity and a positive smoking history would also be at increased BE risk and would equally meet eligibility criteria.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of prior EGD procedure in past ten years
* Inability to provide written informed consent
* History of weekly of more frequent heartburn or regurgitation for five or more years
* On anti-coagulant drug(s) that cannot be temporarily discontinued or coagulopathy with INR > 1.5
* Known history of esophageal varices or esophageal stricture
* Any contraindication, as deemed in Investigator's medical judgment, to undergoing the EsoCheck procedure, undergoing the EGD procedure, and/or having biopsies taken, including but not limited to due to comorbidities such as coagulopathy or a known history of esophageal diverticula, esophageal fistula and/or esophageal ulceration
* History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills
* Oropharyngeal tumor
* History of esophageal or gastric surgery, with exception of uncomplicated surgical fundoplication procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-09-27 (Estimated); Study Completion 2029-09-27 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value for Barret's Esophagus in EsoCheck/EsoGuard positive participants | Up to 5 years
  The primary goal of this study is to develop a non-endoscopic screening test for the non-GERD population that provides a PPV >20%, i.e. at least 2-fold greater than the 10% PPV of society recommended EGD screening of chronic GERD patients with any additional risk factors.
Barrett's Esophagus prevalence in EsoCheck/EsoGuard test negative subjects from a high-risk GERD negative population | Up to 5 years
  This study will also perform endoscopy in a sample of EC/EG negative subjects to confirm that BE is enriched in the test positive versus test negative population. This will be measured by the prevalence of BE in a high-risk GERD negative population.
Tissue origins of true positive versus false positive EsoCheck/EsoGuard tests in non-GERD screening population | Up to 5 years
  In BE positive cases, biopsies will be taken every 2-cm across the BE segment to map the extent of the field of methylated Vimentin (mVim) and methylated CCNA1 (mCCNA1) DNA detected by EsoGuard.

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Chak, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No